CLINICAL TRIAL: NCT02096523
Title: Use of Proteomics for the Diagnosis of a Platelet-related Bleeding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ela Shai (Other)
Responsible Party: Sponsor-Investigator, Ela Shai, Researcher at Hadassah Medical Center, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 002714- HMO-CTIL
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Inherited Platelet Disorders
Keywords: inherited platelet disorders; proteome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet disease (Experimental): patients with inherited platelet disorders
  Interventions: Other: Blood collection for platelet protein samples
- Healthy (Experimental): Healthy family members of patients with inherited platelet disorders
  Interventions: Other: Blood collection for platelet protein samples

INTERVENTIONS:
Other: Blood collection for platelet protein samples

SUMMARY:
The goal of this study is to identify the platelet defect responsible for the bleeding in families from our inherited platelet disorders Israeli-Palestinian registry. The investigators plan to characterize platelet proteome expression after removing high abundance proteins. The investigators will compare the proteome of sick and healthy members of families with inherited platelet disorders, and identify and validate structural proteins, signaling cascades and biomarkers for detection and diagnosis of unknown platelet disorders. The investigators expect to discover new key findings that allow better understanding of human platelet function and allow better diagnosis and treatment of patients with inherited platelet function disorders.

ELIGIBILITY:
Inclusion Criteria:

* History of inherited platelet disorders in the family

Exclusion Criteria:

* none

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Levels of detectable platelet proteins | 2014-2015 (1 year)
  Characterize platelet proteome expression profile

SECONDARY OUTCOMES:
Changes in protein expression from sick and healthy platelets | 2015-2019 (4 years)
  Analysis of platelet proteome of sick and healthy members of families with inherited platelet disorders

OTHER OUTCOMES:
Number of proteins that inducate disease | 2017-2019 (2 years)
  Identify and validate a panel of specific biomarkers candidates

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel